CLINICAL TRIAL: NCT02476422
Title: A Randomized, Double-blind, Double-dummy, Active-controlled Study to Assess the Efficacy and Tolerability of 50 mg Diclofenac Potassium Soft Gelatin Capsules Compared With 400 mg Ibuprofen Tablets in Patients With Moderate to Severe Postoperative Dental Pain
Brief Title: A Study to Assess the Efficacy and Tolerability of Diclofenac Potassium Soft Gelatin Capsules Compared With Ibuprofen Tablets in Patients With Moderate to Severe Postoperative Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCAT458M2402
Record Dates: First submitted 2015-05-18; First posted 2015-06-19 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Post Operative Dental Pain
Keywords: Diclofenac potassium; Post-operative dental pain; Moderate to severe pain
MeSH Terms: interventions — Diclofenac; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dilcofenac potassium + placebo to Ibuprofen (Experimental): Single dose of diclofenac potassium 50 mg soft gelatin capsule was given once patient developed moderate to severe pain post the extraction of two ipsilateral third molar teeth. Single dose of placebo to ibuprofen 400 mg tablet was also given to patient in order to maintain double dummy method.
  Interventions: Drug: Diclofenac potassium; Drug: Placebo to ibuprofen
- Ibuprofen + placebo to diclofenac potassium (Active Comparator): Single dose of ibuprofen 400 mg tablet was given once patient develops moderate to severe pain post the extraction of two ipsilateral third molar teeth. Single dose of placebo to diclofenac potassium 50 mg soft gelatin capsule was also given to patient in order to maintain double dummy method.
  Interventions: Drug: Ibuprofen; Drug: Placebo to diclofenac potassium

INTERVENTIONS:
Drug: Diclofenac potassium — Single dose of diclofenac 50 mg soft gelatin capsule
  Other Names: diclofenac-K
  Arms: Dilcofenac potassium + placebo to Ibuprofen
Drug: Ibuprofen — Single dose of ibuprofen 400 mg tablet
  Other Names: Ibuprofen acid
  Arms: Ibuprofen + placebo to diclofenac potassium
Drug: Placebo to ibuprofen — Single dose of placebo to ibuprofen 400 mg tablet
  Other Names: Placebo
  Arms: Dilcofenac potassium + placebo to Ibuprofen
Drug: Placebo to diclofenac potassium — Single dose of placebo to diclofenac potassium 50 mg soft gelatin capsule
  Other Names: Placebo
  Arms: Ibuprofen + placebo to diclofenac potassium

SUMMARY:
The study is designed to assess the efficacy and tolerability of diclofenac potassium soft gelatin capsules compared with ibuprofen tablets in patients with moderate to severe postoperative dental pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients requiring surgical removal of 2 ipsilateral third molars, of which the mandibular must be fully or partially impacted. The ipsilateral maxillary third molar may be of any impaction level.
* Patients having a moderate to severe Baseline pain intensity as assessed by a score of 2 (moderate) or 3 (severe) on the 4-point categorical pain intensity VRS, confirmed by a VASPI score of ≥ 50 mm within 5 hours of surgical completion, after local anesthetic dissipation.

Key Exclusion Criteria:

* Patients who require the removal of a single third molar, or 2 ipsilateral third molars where mandibular molar is not fully or partially impacted.
* Patients with active peptic ulcer disease or a history of significant gastrointestinal disease or any gastrointestinal bleeding.
* Patients with coagulation or bleeding disorders.
* Patients with a positive drug or alcohol screen.
* Patients who have received an anti-inflammatory agent, analgesic, sedative, hypnotic, muscle relaxant, or tranquilizer within 5 elimination half-lives before administration of study drug (other than surgical anesthetic prior to and during dental surgery).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Started | 166 ("started" = Randomized Set/Full analysis set/Safety set) | 162
Completed | 166 | 161
Not Completed | 0 | 1
Not completed — Subject/guardian decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set included all subjects who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium | Total
Number analyzed (Participants) | 166 | 162 | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.9 (5.21) | 24.7 (6.11) | 24.8 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 96 | 194
  Male | 68 | 66 | 134

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analog Scale of Pain Intensity (VASPI) at 60 Minutes Post Dose
Description: VASPI reduction from baseline is the difference between the Baseline VASPI score and the VASPI score at a specific observation point. Subjects were asked to identify their current level of pain intensity on the 100 mm VASPI, labeled "no pain" (0 mm) as the left anchor and "worst possible pain" (100 mm) as the right anchor. A positive change represents a reduction in pain.
Time Frame: 60 minutes postdose
Population: The efficacy analyses were performed on the full analysis set (FAS) which consisted of all randomized subjects who were exposed to study drug and provided at least 1 post-dose assessment on any efficacy parameter. Last observation carried forward (LOCF) was used as the imputation technique.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
units on a scale | 47.3 (2.06) | 44.1 (2.08)
Statistical Analysis 1: Comparison: Dilcofenac Potassium + Placebo to Ibuprofen vs Ibuprofen + Placebo to Diclofenac Potassium; Test type: Superiority or Other; p = 0.211, ANCOVA; Mean Difference (Net) = 3.2, 95% CI 2-sided [-1.8 to 8.3]

2. Secondary Outcome: Change From Baseline in Visual Analog Scale of Pain Intensity (VASPI) at Different Time Points
Description: as for outcome 1
Time Frame: 15, 30, 45, and 90 minutes, and 2, 4, 5, 6, 7, and 8 hours post dose
Population: The efficacy analyses were performed on the full analysis set (FAS), which consisted of all randomized subjects who were exposed to study drug and provided at least 1 post-dose assessment on any efficacy parameter. Last observation carried forward (LOCF) was used as the imputation technique.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
Units on a scale
  15 minutes | 9.2 (1.55) | 13.7 (1.56)
  30 minutes | 24.1 (1.96) | 26.6 (1.98)
  45 minutes | 38.9 (2.16) | 36.7 (2.18)
  90 minutes | 53.5 (1.98) | 49.1 (2.00)
  2 hours | 55.6 (1.96) | 53.0 (1.98)
  4 hours | 48.8 (2.22) | 51.9 (2.24)
  5 hours | 45.4 (2.40) | 49.8 (2.42)
  6 hours | 40.3 (2.58) | 46.5 (2.61)
  7 hours | 35.2 (2.68) | 41.9 (2.71)
  8 hours | 32.3 (2.74) | 37.7 (2.76)

3. Secondary Outcome: Area Under the Curve (AUC) of Visual Analog Scale of Pain Intensity (VASPI) Measuring Change From Baseline at Different Time Points
Description: VASPI reduction from baseline is the difference between the Baseline VASPI score and the VASPI score at a specific observation point. Subjects were asked to identify their pain intensity using the 100 mm VASPI to indicate their current level of pain intensity on the 100 mm VASPI labeled "no pain" (0 mm) as the left anchor and "worst possible pain" (100 mm) as the right anchor. A positive change shows reduction in pain.
  AUC of VASPI reduction from baseline for each time point was calculated using the trapezoidal rule.
Time Frame: 15, 30, 45, 60 and 90 minutes, and 2, 4, 5, 6, 7, and 8 hours post dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale*hours
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
units on a scale*hours
  15 minutes | 16.1914 (0.19369) | 15.6262 (0.19558)
  30 minutes | 29.3759 (0.58537) | 27.9216 (0.59109)
  45 minutes | 38.8570 (1.03408) | 37.3448 (1.04418)
  60 minutes | 45.4321 (1.48887) | 44.5882 (1.50342)
  90 minutes | 54.9330 (2.34986) | 55.9885 (2.37282)
  2 hours | 62.3674 (3.15839) | 65.1654 (3.18925)
  4 hours | 96.7669 (6.56154) | 98.9982 (6.62565)
  5 hours | 119.0564 (8.50377) | 117.4797 (8.58686)
  6 hours | 145.6112 (10.58291) | 138.6947 (10.68631)
  7 hours | 177.2751 (12.76115) | 163.8821 (12.88584)
  8 hours | 212.9300 (15.01237) | 193.4450 (15.15905)

4. Secondary Outcome: Time to Confirmed First Perceptible Pain Relief
Description: Time to onset of first perceptible pain relief (FPR), provided the FPR was subsequently 'confirmed' through the achievement of meaningful pain relief (MPR). Participant started two stopwatches at dosing, and recorded FPR by stopping the first stopwatch when he/she first experienced 'any' pain relief. FPR is 'confirmed' only if the participant also stopped the second stopwatch indicating 'meaningful pain relief'.
Time Frame: Within 8 hours postdose
Population: The efficacy analyses were performed on the full analysis set (FAS), which consisted of all randomized subjects who were exposed to study drug and provided at least 1 postdose assessment on any efficacy parameter.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
minutes | 15.81665 [11.55000 to 29.13330] | 14.98335 [9.88330 to 22.16670]

5. Secondary Outcome: Time to Onset of Meaningful Pain Relief (MPR)
Description: Using the double stopwatch technique, participant started two stopwatches at dosing, and stopped the second stopwatch as soon as he/she began to experience 'meaningful' relief from pain. Time elapsed is recorded as the MPR.
Time Frame: Within 8 hours postdose
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
minutes | 41.67500 [29.46670 to 60.11670] | 42.02500 [24.90000 to 73.40000]

6. Secondary Outcome: Time to Onset of First Perceptible Pain Relief (FPR)
Description: Using the double stopwatch technique, participant started two stopwatches at dosing, and stopped the first stopwatch as soon as he/she first began to feel 'any' relief from pain. The time elapsed was recorded as the FPR.
Time Frame: Within 8 hours postdose
Population: The efficacy analyses were performed on the full analysis set (FAS), which consisted of all randomized subjects who were exposed to study drug and provided at least 1 post-dose assessment on any efficacy parameter.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
minutes | 15.81665 [11.55000 to 29.13330] | 14.85000 [9.66670 to 21.33330]

7. Secondary Outcome: Sum of Pain Intensity Difference (SPID)
Description: At baseline and at each defined study time point, the clinical site staff captured pain intensity information from each subject using the 4-point categorical VRS. The subject was asked "What is your pain level at this time?" and the response was recorded as 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Pain intensity difference (PID) was the difference between the baseline pain intensity score and the pain intensity score at a specific observation point. SPID is the weighted sum of PIDs from the 15-minute to the 8-hour observation point (SPID8). Additionally, SPID evaluations were also be done at 1 (SPID1), 2 (SPID2), 4 (SPID4) and 6 (SPID6) hours post dose. The weights used for these values were 0.25 for the 15-, 30-, 45-, and 60-minute observations, and 0.5 for the 90-minute, 2- and 4-hour observations, and 1 for the remaining observations.
Time Frame: 1, 2, 4, 6, and 8 hours postdose
Population: The efficacy analyses were performed on the full analysis set (FAS), which consisted of all randomized subjects who were exposed to study drug and provided at least 1 postdose assessment on any efficacy parameter. Last observation carried forward (LOCF) was used as the imputation technique.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
units on a scale
  SPID1 | 1.077 (0.0525) | 1.049 (0.0530)
  SPID2 | 2.955 (0.1050) | 2.772 (0.1060)
  SPID4 | 6.165 (0.2276) | 6.196 (0.2298)
  SPID6 | 8.970 (0.3703) | 9.323 (0.3739)
  SPID8 | 11.099 (0.5180) | 11.904 (0.5230)

8. Secondary Outcome: Summed Total Pain Relief (TOTPAR) at Different Time Points
Description: After the administration of the single dose of the assigned study treatment, at the defined study time points, the clinical site staff captured pain relief information from each subject.
  The subject was asked "What is the amount of pain relief as compared to the starting pain?" and the response was recorded as 0 = none, 1 = a little, 2 = some, 3 = a lot, or 4 = complete.
  Total pain relief (TOTPAR) was the weighted sum of the pain relief scores from the 15-minute to the 8-hour observation points (TOTPAR8). Additionally, TOTPARs at 1, 2, 4 and 6 hours were calculated. The weights used for these values (evaluation time points) were 0.25 for the 15-, 30-, 45-, and 60-minute observations, 0.5 for the 90-minute, 2- and 4-hour observations, and 1 for the remaining observations.
Time Frame: 1, 2, 4, 6, and 8 hours postdose
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
units on a scale
  TOTPAR1 | 1.807 (0.0680) | 1.780 (0.0687)
  TOTPAR2 | 5.032 (0.1452) | 4.817 (0.1466)
  TOTPAR4 | 10.642 (0.3353) | 10.848 (0.3385)
  TOTPAR6 | 15.647 (0.5595) | 16.499 (0.5650)
  TOTPAR8 | 19.679 (0.7915) | 21.341 (0.7992)

9. Secondary Outcome: Peak Analgesic Effect
Description: Peak analgesic relief is represented through highest pain intensity difference (PID), highest VASPI reduction, and highest pain relief scores. Pain intensity was measured on a verbal rating scale (VRS) ranging from 0 to 3 (none to severe, with higher score for higher pain intensity). PID represents difference in this score at baseline and specific time points, larger change indicating larger reduction in pain, with highest PID representing the largest difference. Pain relief was recorded on a scale ranging from 0 to 4 (none to complete, with higher score for higher pain relief), with highest pain relief representing maximum relief obtained. Pain intensity was also measured through a 100 mm visual analogue scale (VASPI), ranging from "no pain" (0 mm) to "worst possible pain" (100 mm). A positive change in VASPI indicates reduction in pain, with highest VASPI reduction representing highest change.
Time Frame: From dose administration to 8 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
units on a scale
  Highest Mean PID | 1.9 (0.72) | 1.8 (0.74)
  Highest pain relief | 3.6 (0.74) | 3.5 (0.86)
  Highest VASPI reduction | 61.3 (17.99) | 60.2 (19.35)

10. Secondary Outcome: Duration of Analgesia
Description: Duration of analgesia (time to first use of rescue medication) was evaluated, from dose administration to the time of first use of rescue medication within the 8-hour treatment period. Censored observations were included in calculating this endpoint. Censored subjects include any subject who did not take rescue medication prior to the end of the assessment period of 480 minutes (8 hours).
Time Frame: From dose administration to 8 hours post dose
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
minutes | 480.0 [383.0 to 480.0] | 480.0 [480.0 to 480.0]

11. Secondary Outcome: Number of Patients Needing Rescue Medication
Description: The number of patients needing rescue medication within the 8 hour treatment period was evaluated.
Time Frame: From dose administration to 8 hours post dose
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
Participants | 47 | 36

12. Secondary Outcome: Number of Patients With Different Responses Based on Patient's Global Assessment of Response to Treatment (PGART)
Description: PGART was measured by asking patients to give a score on a scale from 0 to 4, where 0 = poor; 1 = fair; 2 = good; 3 = very good; 4 = excellent. This measurement was taken at the end of 8 hours, or before the use of rescue medication (for a patient who takes rescue medciation within the 8 hour period).
Time Frame: At 8 hour postdose prior to use of rescue medication
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
Participants
  Poor (0) | 6 | 10
  Fair (1) | 7 | 7
  Good (2) | 49 | 34
  Very good (3) | 55 | 64
  Excellent (4) | 49 | 47

13. Secondary Outcome: Number of Patients With Any Adverse Events, Serious Adverse Events and Death
Description: Treatment emergent adverse events are reported in the below data table.
Time Frame: time of dosage administration up to the follow-up phone call on study Day 3 (maximum 3 days)
Population: Safety analyses were performed on the safety set, which included all randomized subjects who were exposed to study drug.
Measure: Number; unit: Participants
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Number analyzed (Participants) | 166 | 162
Participants
  any adverse events | 47 | 47
  serious adverse events | 0 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Time of dosage administration up to the follow-up phone call on study Day 3 (maximum 3 days)
Description: The safety set consisted of all randomized subjects who were exposed to study drug. Treatment emergent adverse events are reported.
Arm/Group | Dilcofenac Potassium + Placebo to Ibuprofen | Ibuprofen + Placebo to Diclofenac Potassium
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/162
Other Adverse Events (participants affected / at risk) | 47/166 | 47/162
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dilcofenac Potassium + Placebo to Ibuprofen (N=166) | Ibuprofen + Placebo to Diclofenac Potassium (N=162)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 10
Vomiting (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 10 | 5
Headache (Nervous system disorders) | 27 | 33
Hypoaesthesia (Nervous system disorders) | 5 | 5
Syncope (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.